CLINICAL TRIAL: NCT00691184
Title: A Double-Blind, Randomized, Parallel Design Study To Assess the Safety and Pharmacokinetics of Terbinafine Hydrogen Cloride (HCl) Nail Lacquer Applied for 28 Days in Patients With Onychomycosis
Brief Title: Safety and Pharmacokinetics of Terbinafine Hydrogen Chloride (HCl) Nail Lacquer in Patients With Onychomycosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NexMed (U.S.A.), Inc. (subsidiary of Apricus Biosciences, Inc.) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NM-060-1001
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Onychomycosis/Onycholysis and Tinea Pedis
Keywords: Onychomycosis, Toenail fungal infection, Terbinafine HCl, Pharmacokinetics
MeSH Terms: conditions — Onychomycosis; Onycholysis; Tinea Pedis | interventions — Terbinafine; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Group 1 (Experimental): 0% Terbinafine HCl Nail Lacquer for 28 days.
  Interventions: Drug: Placebo
- Group 2 (Experimental): 10% Terbinafine HCl Nail Lacquer.
  Interventions: Drug: Terbinafine Hydrochloride
- Group 3 (Active Comparator): 1% Lamisil® Cream
  Interventions: Drug: Terbinafine Hydrochloride
- Group 4 (Active Comparator): Dose of 250 mg Lamisil® Tablets (Groups 1,2,3) at end of study.
  Interventions: Drug: Terbinafine

INTERVENTIONS:
Drug: Placebo — 0% Terbinafine HCl Nail Lacquer for onychomycosis, twice daily for 28 days.
  Arms: Group 1
Drug: Terbinafine Hydrochloride — 10% Terbinafine HCl Nail Lacquer for onychomycosis, twice daily for 28 days.
  Arms: Group 2
Drug: Terbinafine Hydrochloride — 1% Terbinafine Hydrochloride Cream, twice a day for 7 days.
  Other Names: Lamisil® Cream, 1%
  Arms: Group 3
Drug: Terbinafine — Terbinafine tablet, 250mg, single dose in groups 1,2 and 3 at end of study.
  Other Names: Lamisil, 250mg tablet
  Arms: Group 4

SUMMARY:
In this study, the safety and pharmacokinetics of 10 % terbinafine hydrogen chloride (HCl) nail lacquer wre investigated by comparison with vehicle control and 1% terbinafine cream

DETAILED DESCRIPTION:
This was a double-blind, randomized, parallel-design, placebo-controlled Phase 1 study comparing 10% Terbinafine HCl Nail Lacquer vs. Placebo Nail Lacquer (i.e., vehicle control). For comparative purposes, the study also included a contemporaneous assessment of 1% Lamisil® Cream (1% terbinafine HCl) and Lamisil® Tablets (terbinafine HCl labeled as 250 mg of terbinafine).

Forty (40) onychomycosis (Groups 1 and 2) and 16 tinea pedis (Group 3) patients were enrolled at 3 study centers. In Group 1, 10% Terbinafine HCl Nail Lacquer, and, in Group 2, its vehicle (0% terbinafine HCl), were applied topically by brushing on a dose volume of approximately 10 μL per nail twice daily for 28 days to each toenail and to 5 mm of adjacent skin. The patients visited the study center on Days 3, 7, 14, 21, and 28 for assessments of clinical signs and to obtain blood samples. In addition, a 24-hour urine sample was collected and assessed on Day 28 and Day 35. Fifty six (56) patients (20 in Group 1, 20 in Group 2, and 16 in Group 3) received a single oral dose of a 250 mg Lamisil® Tablet after a 7-day washout period.

For comparative purposes, the study also evaluated the local and systemic safety, and plasma levels of terbinafine, and its 3 major metabolites (i.e., desmethyl terbinafine, carboxybutyl terbinafine, and desmethyl carboxybutyl terbinafine) following administration of 1% Lamisil® Cream in comparison with 10% Terbinafine HCl Nail Lacquer. In Group 3, approximately 0.5 g of 1% Lamisil® Cream was applied twice a day for 7 days to the area of the foot affected with tinea pedis. The patients visited the study center on Day 3 and on Day 7 for assessments of clinical signs and collection of blood samples. A 24-hour urine sample was collected and assessed on Day 7 and Day 14.

ELIGIBILITY:
Inclusion Criteria:

Patients were required to meet all of the following criteria in order to be eligible for entry in the study:

* Were between 18 and 70 years of age, of any race and of either sex;
* Were in good general health as confirmed by a medical history and brief physical examination;
* Groups 1 and 2, presented with clinically diagnosed stable or exacerbating onychomycosis with more than 25 % involvement of one great toenail;
* For Group 3, had mild tinea pedis (mild tinea pedis was defined as mild erythema, mild scaling, cracking or fissuring, and mild burning or pruritus);
* For Groups 1 and 2, had at least five toenails with onycholysis;
* For Groups 1 and 2, a positive calcofluor (KOH) exam must have been obtained during Visit 1 from specimens taken from the affected great toenail;
* Signed a statement of informed consent;
* Were able to understand the requirements of the study, abide by the restrictions, and return for all of the required examinations;
* If female, met one of the following criteria: (a) had been post-menopausal for at least one year, or (b) had a hysterectomy or tubal ligation, or (c) was using oral/systemic contraceptives or an intrauterine device at least 28 days prior to study entry and throughout the study, or (d) agreed to use spermicide in combination with barrier methods of contraception throughout the study;
* Had 10 toes with nails that could be clipped to provide nail samples.

Exclusion Criteria:

Any of the following excluded a patient from participating in the study:

* Any missing toes;
* Known hypersensitivity to terbinafine or any of the excipients in the nail lacquer;
* Vital signs measurement that were clinically significantly outside the normal limits;
* Liver function test values more than two times the upper limit of normal or other clinical laboratory values, which were clinically significantly outside normal limits;
* Receipt of terbinafine tablets within 12 months or terbinafine cream or solution within six months prior to screening;
* Participation in a clinical trial for the systemic treatment of onychomycosis within the previous two months;
* Current treatment with rifampin, phenobarbital, phenytoin, carbamazepine, terfenadine, or digoxin;
* Prior treatment with an investigational drug within one month prior to study start;
* Diagnosis of psoriasis or history of psoriasis;
* Diagnosis of a serious concurrent disease that might prevent completion of the trial;
* Pregnancy (confirmed by pregnancy test), or plan to become pregnant within the study period or nursing;
* Inability to read, understand, or sign the informed consent form or the patient instructions for applying and removing the study formulations;
* Inability to apply the study medication;
* Onychomycosis patient unwilling to provide nail clippings;
* Inability to provide adequate blood sample;
* Use of any nail polish products or other nail cosmetic products within seven days prior to the start of treatment, or unwilling to discontinue use of these products during the course of this study.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2005-02; Primary Completion 2005-06 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The primary safety objective was to determine the safety of 10% Terbinafine HCl Nail Lacquer by assessing local and systemic adverse experiences, changes in vital signs, clinical laboratory test results, physical examinations, and electrocardiogram (ECG) | 28 Days

SECONDARY OUTCOMES:
To determine plasma levels of terbinafine and its metabolites after administration of 10% Terbinafine HCl Nail Lacquer to toenails, 1% Lamisil® Cream to the infected (i.e., tinea pedis) area of the foot and a single Lamisil® Tablet (250 mg) on Day 35. | 3, 7, 14, 21 and 28 days and Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Ming Q Lu, MD., Ph.D., Study Director — NexMed (U.S.A.), Inc.
Locations (1):
- TKL Research Inc., Paramus, New Jersey, United States